CLINICAL TRIAL: NCT07402980
Title: Polycystic Ovary Syndrome Symptoms Inventory: Development, Validity and Reliability in Turkey
Brief Title: Development of the Polycystic Ovary Syndrome Symptoms Inventory
Status: Recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Büşra Boğa, Research Assistant, Abant Izzet Baysal University
Other Study IDs: AIBU-HEM-BB-01
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Polycystic Ovary Syndrome; Psychological Distress
Keywords: Polycystic Ovary Syndrome; Symptom Burden; Psychological Distress; Inventory Development
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women diagnosed with PCOS: Women aged 18-49 who report having been diagnosed with PCOS will be included in the study.

SUMMARY:
Polycystic Ovary Syndrome Symptom Severity and Distress Inventory: Development, Validity and Reliability in Turkey

The goal of this observational study is to develop and validate a self-report inventory that assesses Polycystic Ovary Syndrome (PCOS) symptoms and the level of distress experienced by women diagnosed with PCOS. The main question it aims to answer is:

Is the newly developed inventory a valid and reliable instrument for assessing PCOS symptoms and related distress in women?

Participants will answer online survey questions including a demographic information form and three scales evaluating psychological health and PCOS related symptoms, including the newly developed symptom and distress inventory.

DETAILED DESCRIPTION:
The research is a methodological scale development study.

A review of the literature reveals that despite strong evidence linking Polycystic Ovary Syndrome (PCOS) to anxiety, depression, and diminished quality of life, current assessment tools often fail to adequately represent psychological symptoms. There is a critical need for holistic and culturally sensitive instruments that address both the physical and psychological dimensions of PCOS. It is therefore thought that the developed scale will fill an important gap.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman aged 18-49 (of reproductive age) who states she has been diagnosed with PCOS
* Being able to read and understand Turkish
* Volunteering to participate in the study

Exclusion Criteria:

* Having a disease that could cause symptoms similar to PCOS (such as Cushing's syndrome, thyroid dysfunction, hyperprolactinemia, androgen-secreting tumors)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of women aged 18-49 who have been diagnosed with Polycystic Ovary Syndrome (PCOS). The study aims to reach a sample size of at least 85 to 170 participants. Women who meet the inclusion criteria and agree to participate on a voluntary basis will be invited to the study.
  Data will be collected via an online survey form prepared by the researchers. Participants will be recruited through social media platforms (such as WhatsApp and Instagram). To ensure ethical standards, an informed consent text will be included at the beginning of the online form, and a mandatory question will be used to confirm voluntary participation. Additionally, a mandatory screening question regarding PCOS diagnosis will be included to verify that participants meet the inclusion criteria; individuals without a PCOS diagnosis will be excluded from the sample.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Polycystic Ovary Syndrome Symptom Severity and Distress Inventory | At the time of survey completion (Baseline)
  The newly developed inventory consists of 34 items in total, with 17 items dedicated to evaluating PCOS symptom severity and 17 items for measuring distress levels. Each item is scored on a scale from 0 to 10. Total scores are calculated separately for symptom severity and distress levels, with each score ranging from 0 to 100. Higher scores on these measurements indicate an increase in both symptom severity and the level of distress experienced by the participant.

SECONDARY OUTCOMES:
Participant Information Form | At the time of survey completion (Baseline)
  A 10-item form developed by the researchers to collect sociodemographic data, such as age and educational background, as well as specific questions regarding the participants' Polycystic Ovary Syndrome (PCOS) history.
Health-Related Quality of Life Questionnaire-50 for Polycystic Ovary Syndrome (PCOSQ-50) | At the time of survey completion (Baseline)
  This scale is designed to determine the impact of Polycystic Ovary Syndrome (PCOS) on quality of life. It consists of 50 items and 6 subscales: psychosocial and emotional, fertility, sexual function, obesity and menstrual disorders, hirsutism, and coping. Total scores range from 50 to 250. Subscale scores are determined by calculating the average score of the items answered within that specific domain. Unanswered items are excluded from the average score calculation.
Kessler Psychological Distress Scale (K10-PDS) | At the time of survey completion (Baseline)
  This 10-item scale measures the frequency of symptoms such as nervousness, hopelessness, sadness, worthlessness, and fatigue to assess non-specific psychological distress. The scale is a 5-point Likert-type instrument, with total scores ranging from 10 to 50. Higher scores indicate higher levels of psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Melisa Bulut, PhD, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect the confidentiality and privacy of the participants.